CLINICAL TRIAL: NCT07039812
Title: The Effect of Virtual Reality and Eye Mask Application During Dressing After Coronary Artery Bypass Graft Surgery on Sternotomy Pain, Anxiety, and Physiological Parameters
Brief Title: The Effect of Virtual Reality and Eye Mask During Dressing After CABG Surgery
Acronym: CABG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Tugce Bozkurt Elmas, PhD Candidate, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CABG-15
Record Dates: First submitted 2025-06-03; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: CABG; Physiological Parameter; Postoperative Pain; Postoperative Anxiety; Coronary Artery Disease
Keywords: Coronary Artery Bypass Graft; Virtual Reality; Eye Mask; Pain Management; Anxiety; Physiological Parameter
MeSH Terms: conditions — Pain, Postoperative; Coronary Artery Disease; Agnosia; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three parallel arms: VR intervention, eye mask intervention, or standard care control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual Reality Group (Experimental): Participants in this group will watch 360-degree nature-themed videos through a virtual reality headset (Oculus meta quest 2) during both the first and second sternotomy dressing procedures.
  Interventions: Device: Virtual Reality Headset
- Eye Mask Group (Experimental): Participants in this group will wear an eye mask during both the first and second sternotomy dressing procedures.
  Interventions: Device: Eye Mask
- Control Group (No Intervention): Participants in this group will receive standard postoperative care during dressing, with no additional interventions applied.

INTERVENTIONS:
Device: Virtual Reality Headset — During the dressing change, nature-themed videos will be shown through a virtual reality headset that immerses the user in a 360-degree, three-dimensional virtual environment.
  Arms: Virtual Reality Group
Device: Eye Mask — A soft, adjustable, 3D-structured eye mask (Poblex brand) will be applied during the dressing procedure.
  Arms: Eye Mask Group

SUMMARY:
This study aims to evaluate the effects of virtual reality (VR) and eye mask (EM) applications on pain, anxiety, and physiological parameters during dressing after Coronary Artery Bypass Graft (CABG) surgery.

Postoperative dressing procedures, especially after sternotomy, often cause significant pain and anxiety in patients. These issues can negatively impact recovery and increase the need for medication. Non-pharmacological interventions such as VR and EM may help reduce these symptoms.

In this randomized controlled trial, 90 patients are divided into three groups: VR group, EM group, and a control group receiving standard care. Pain and anxiety levels are monitored baseline, immediately after, and 15 minutes after both the first and second dressing procedures. Physiological parameters are measured baseline, during, immediately after, and 15 minutes after both dressing procedures. Additionally, analgesic use is followed baseline and immediately after each dressing procedure. The study is conducted in a cardiovascular intensive care unit in Istanbul, Türkiye. It is expected that the findings will support the integration of VR and EM as effective, low-cost, and non-invasive options for postoperative care, improving patient comfort and healthcare quality.

DETAILED DESCRIPTION:
This randomized controlled experimental study investigates the effects of virtual reality (VR) and eye mask (EM) applications on sternotomy pain, anxiety, and physiological parameters during postoperative dressing following Coronary Artery Bypass Graft (CABG) surgery.Pain and anxiety during dressing procedures after CABG surgery can negatively affect the recovery process, increase stress responses, prolong hospital stays, and raise the need for medication. Non-pharmacological interventions such as VR and EM are considered effective strategies for managing these symptoms.

The study includes 90 patients, randomly assigned to one of three groups: VR Group: Patients watched 360-degree nature-themed videos using a virtual reality headset during dressing. EM Group: Patients wore an eye mask during dressing. Control Group: Patients received standard care without any additional intervention. The study is being conducted in the Cardiovascular Surgery Intensive Care Unit of a public hospital located in Istanbul, Türkiye.

Inclusion criteria include adult patients undergoing CABG for the first time, ASA classification I-II-III, fully conscious, oriented, cooperative, and willing to provide informed consent. Exclusion criteria include patients with infections or complications, psychiatric disorders, or sensory impairments such as hearing or vision problems. Pain and anxiety levels are assessed at three time points during both the first and second dressing procedures: baseline, immediately after dressing, and 15 minutes after dressing. Physiological parameters (blood pressure, pulse rate, respiratory rate, oxygen saturation) are measured at four time points: baseline, immediately after dressing, and 15 minutes after dressing. Analgesic use is recorded baseline and immediately after each dressing. This study is one of the first to compare VR and EM interventions in the context of high-risk, postoperative cardiac surgery. The results are expected to contribute to evidence-based nursing practices, improve patient comfort in the postoperative period, and support the use of cost-effective, drug-free alternatives for pain and anxiety management in clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years
* First-time coronary artery bypass graft (CABG) surgery for coronary artery disease
* ASA physical status I, II, or III
* Conscious, oriented, and cooperative
* Able to communicate verbally
* Provided written informed consent

Exclusion Criteria:

* Presence of sternal wound infection or inflammation
* Intubated at the time of assessment
* Undergoing revision surgery
* Receiving anesthesia or sedation in the ICU
* Experiencing intraoperative or postoperative complications
* Inability to speak Turkish
* Hearing or visual impairment
* Diagnosed psychiatric or cognitive disorder
* Diagnosis of epilepsy
* Body mass index (BMI) ≥ 30
* Participation in another clinical trial during the same period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | Baseline, immediately after, and 15 minutes after first and second dressing
  Pain intensity will be measured using the Visual Analog Scale (VAS) at three time points: before, immediately after, and 15 minutes after both the first and second sternotomy dressing procedures.
State-Trait Anxiety Inventory (STAI-II) | Baseline, immediately after, and 15 minutes after first and second dressing
  State anxiety levels (STAI-I) will be measured before, immediately after, and 15 minutes after both the first and second dressing procedures. Trait anxiety (STAI-II) will be measured only once, before surgery.

SECONDARY OUTCOMES:
Physiological Parameters (Blood pressure) | Baseline, during, immediately after, and 15 minutes after first and second dressing
  Blood pressure will be monitored using a monitor device.
Physiological Parameters (Pulse) | Baseline, during, immediately after, and 15 minutes after first and second dressing
  Pulse will be monitored using a monitoring device.
Physiological Parameters (SpO₂) | Baseline, during, immediately after, and 15 minutes after first and second dressing
  Saturation values will be monitored using a monitoring device.
Physiological Parameters (Respiratory rate ) | Baseline, during, immediately after, and 15 minutes after first and second dressing
  Respiratory rate will be monitored using a monitoring device.

OTHER OUTCOMES:
Analgesic Use Frequency | Baseline and immediately after first and second dressing
  Analgesic agents administered in the intensive care unit, including their names, routes of administration, dosages, and timing, will be systematically documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Dr. Cemil Taşçıoğlu City Hospital, Istanbul, Marmara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No